CLINICAL TRIAL: NCT00744848
Title: Phase 3, Multicenter, Randomized, Double-Blind, Parallel-group, Active-control Study to Evaluate the Safety and Efficacy of a Single Administration of SKY0402 for Prolonged Postoperative Analgesia in Subjects Undergoing Hemorrhoidectomy
Brief Title: Study to Evaluate Postoperative Analgesia in Subjects Undergoing Hemorrhoidectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SIMPLE Hemorrhoidectomy 312
Record Dates: First submitted 2008-08-28; First posted 2008-09-01 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Hemorrhoids
Keywords: hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine HCl (Active Comparator): 100 mg Bupivacaine HCl (e.g., Marcaine with epinephrine 1:200,000) is the reference-listed drug for bupivacaine and contains the same active, local anesthetic as SKY0402.
  A single dose of study drug was administered intraoperatively (at the end of surgery) via local infiltration.
  Interventions: Drug: Bupivacaine HCl
- SKY0402 (Other): 300 mg SKY0402 in a 40-mL injection volume.
  A single dose of study drug was administered intraoperatively (at the end of surgery) via local infiltration.
  Interventions: Drug: SKY0402

INTERVENTIONS:
Drug: Bupivacaine HCl — 100 mg Bupivacaine HCl
  Other Names: Marcaine with epinephrine 1:200,000
  Arms: Bupivacaine HCl
Drug: SKY0402 — Single administration 300 mg SKY0402 in a 40-mL injection volume
  Other Names: DepoBupivacaine
  Arms: SKY0402

SUMMARY:
Effective postoperative pain control to promote improved healing, faster patient mobilization, shortened hospital stays, and reduced healthcare costs.

DETAILED DESCRIPTION:
Effective postoperative pain control is a critical element in patient recovery, as the majority of patients may experience significant pain, particularly in the first few days following surgery. Appropriate postoperative pain management contributes to improved healing, faster patient mobilization, shortened hospital stays, and reduced healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female equal or greater than 18 years of age at Screening
* Female subjects: postmenopausal, surgically sterile, or willing to use acceptable means of contraception for at least 30 days after surgery, nonheterosexual lifestyle, or strictly monogamous relationship with a partner who has had a vasectomy.
* Scheduled to undergo 2-or3-column excisional hemorrhoidectomy
* American Society of Anesthesiology (ASA) Physical Class 1-4
* Able and willing to complete with all study visits and procedures
* Able to speak, read, and understand the language of all study forms and instruments used for collecting subject-reported outcomes to provide accurate study assessments
* Willing and capable of provide written informed consent.

Exclusion Criteria:

* Pregnant, nursing or planning to become pregnant during the study period
* Use of any long-acting opioid medication within 3 days of surgery or any opioid medication with 24 hours of surgery.
* Concurrent painful physical condition or concurrent surgery that may require analgesic treatment in the postoperative period for pain not strictly related to the procedure or that may interfere with study assessments.
* Single-column hemorrhoidectomy
* Body weight less than 50 kg (110 pounds)
* History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics, opioid medication, or any ingredient of the medications administered in this study (e.g., sulfites in Marcaine with epinephrine)
* contraindication to epinephrine
* contraindication to any of the pain-control agents planned for postoperative use
* Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug prior to study drug administration
* History of, known addiction, or abuse of illicit drugs, prescription medicines or alcohol within the past 2 years.
* Uncontrolled anxiety schizophrenic, or other psychiatric disorder that may interfere with study assessments or compliance.
* Significant medical conditions or laboratory results that indicate an increased vulnerability to study drugs and procedures, and expose the subject to an unreasonable risk as a result of participating in this clinical trial.
* Any clinically significant event or condition uncovered during surgery
* A cumulative incision length less than 3 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Warnott, RN, ACN-P, Study Director — Pacira Pharmaceuticals, Inc
Locations (20):
- United States (20):
  - West Alabama Research Inc., Birmingham, Alabama
  - Drug Research and Analysis Corporation, Montgomery, Alabama
  - Lotus Clinical Research - Huntington Memorial Hospital, Pasadena, California
  - Accurate Clinical Trials, San Clemente, California
  - UCSD Medical Center, San Diego, California
  - Colon and Rectal Disease Center, Orlando, Florida
  - University of Illinois, Springfield, Illinois
  - Indiana University - Wishard Memorial Hospital, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - CTMG, Inc. - Pitt Medical Center, Greenville, North Carolina
  - Univ. Hospitals of Cleveland, Case Medical Center, Cleveland, Ohio
  - Holston Medical Group, Kingsport, Tennessee
  - Research Concepts, Ltd, Bellaire, Texas
  - Medical Center Ambulatory Surgery Center, Houston, Texas
  - The Women's Hospital of Texas, Houston, Texas
  - Roland Saenz, San Antonio, Texas
  - Multicare Health System, Tacoma, Washington

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine HCl: 100 mg Bupivacaine HCl (e.g., Marcaine with epinephrine 1:200,000) is the reference-listed drug for bupivacaine and contains the same active, local anesthetic as SKY0402.
- SKY0402: Single administration 300 mg SKY0402 in a 40-mL injection volume via local infiltration.
Period: Overall Study
Arm/Group | Bupivacaine HCl | SKY0402
Started | 103 | 101
Completed | 103 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine HCl | SKY0402 | Total
Number analyzed (Participants) | 103 | 101 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 95 | 189
  >=65 years | 9 | 6 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (11.6) | 50.2 (11) | 49.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 48 | 98
  Male | 53 | 53 | 106
Region of Enrollment [Number; unit: participants]
  United States | 103 | 101 | 204

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Numeric Rating Scale at Rest (NRS-R) Pain Intensity Scores
Description: To assess pain intensity at rest (NRS-R), the subject was to assume a resting position that did not exacerbate his or her postoperative pain. The subject was to rest in this position for at least 5 minutes before responding to the following question, "On a scale of 0 to 10, where 0=no pain and 10=worst possible pain, how much pain are you having right now?"
Time Frame: through 96 hours
Population: Note: 204 randomized subjects received study drug and were included in the analyses.
Measure: Mean (Standard Deviation); unit: Units on a scale*hours
Arm/Group | Bupivacaine HCl | SKY0402
Number analyzed (Participants) | 103 | 101
Units on a scale*hours | 359 (194) | 396 (213)

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) Through Day 3 and Serious Adverse Events (SAEs) Through Day 30
Time Frame: through day 30
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bupivacaine HCl | SKY0402
Serious Adverse Events (participants affected / at risk) | 1/103 | 1/101
Other Adverse Events (participants affected / at risk) | 65/103 | 67/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine HCl (N=103) | SKY0402 (N=101)
Chronic Postop Pain (General disorders) | 0 (0) | 1 (1)
Fecal Impaction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine HCl (N=103) | SKY0402 (N=101)
Nausea (Gastrointestinal disorders) | 32 | 38
Constipation (Gastrointestinal disorders) | 12 | 16
Vomiting (Gastrointestinal disorders) | 9 | 16
Flatulence (Gastrointestinal disorders) | 2 | 5
Abdominal Pain (Gastrointestinal disorders) | 0 | 5
Pyrexia (General disorders) | 0 | 8
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 5
Headache (Nervous system disorders) | 7 | 3
Urinary Retention (Renal and urinary disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No